CLINICAL TRIAL: NCT07034170
Title: Comprehensive Interpretation of the Importance of Skeletal Muscle Mass on Prognosis and Recovery in Cardiac Arrest Survivors: From Machine Learning to Clinical Trial
Brief Title: Skeletal Muscle Mass on Prognosis and Recovery in Clinical Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202501085RIND
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Out of Hospital Cardiac Arrest; Inhospital Cardiac Arrest
Keywords: cardiac arrest; Skeletal muscle mass; rehabilitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Intervention Model Description: This is a parallel assignment trial in which participants are allocated to study arms based on the month of admission. Patients admitted during even-numbered months are assigned to the intervention group, while those admitted during odd-numbered months are assigned to the control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- Intervention Group (Experimental)
  Interventions: Behavioral: Enhanced Rehabilitation Program

INTERVENTIONS:
Behavioral: Enhanced Rehabilitation Program — Participants in the intervention group receive an enhanced rehabilitation program, including muscular electrical stimulation, guided active rehabilitation sessions, and structured physical engagement during periods of consciousness. The intervention is designed to promote functional improvement in post-cardiac arrest patients.
  Arms: Intervention Group

SUMMARY:
The objective of this research project is to develop an automated muscle mass measurement system based on computed tomography (CT) images using deep learning and artificial intelligence, and to construct a prognostic prediction model for patients who have experienced cardiac arrest and undergone resuscitation. The model will be validated using multicenter registry data and medical imaging. Furthermore, a clinical trial involving core muscle rehabilitation for post-resuscitation patients will be conducted to evaluate both short-term and long-term outcomes, aiming to comprehensively understand the impact of muscle mass on the prognosis of patients after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic adult patients who experienced sudden cardiac arrest
* Achieved sustained return of spontaneous circulation (ROSC) for more than five minutes following successful resuscitation
* Admitted to the ICU
* Survived beyond 72 hours without successful weaning from mechanical ventilation

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Expected to be weaned from mechanical ventilation within 48 hours
* Terminal-stage cancer or unwillingness to receive aggressive treatment
* Unavailability of ICU care due to overcrowding in the emergency intensive care unit
* Refusal to participate in the study by the patient or family members
* Presence of an implanted pacemaker or defibrillator
* Open wounds, severe edema, or deep vein thrombosis in the lower limbs
* Pre-arrest status limited to wheelchair use or bedridden, unable to ambulate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
skeletal muscle mass | 21 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No